CLINICAL TRIAL: NCT05552924
Title: The Effect of Self Acupressure on Fatigue and Sleep Quality in Epilepsy Patients
Brief Title: Self Acupressure on Fatigue and Sleep Quality in Epilepsy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, gülcan bahcecioğlu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/ 04 - 34
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Epilepsy
Keywords: Self Acupressure; Fatigue; Sleep Quality; Epilepsy Patients
MeSH Terms: conditions — Epilepsy; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Acupressure (Experimental): Each application to the acupressure points (H17, L14, ST36, SP6) will be done in 2 minutes and right and left)
  Interventions: Other: Self-Acupressure
- Control group (No Intervention): Routine maintenance will be applied.

INTERVENTIONS:
Other: Self-Acupressure — Acupressure is a therapy method performed with an instrument or hand, fingertip, palm, elbow, knee, thumb relaxation and wrist bands on various points representing the waist organs in order to ensure the continuation and balance of the energy in our body.
  Arms: Self-Acupressure

SUMMARY:
The aim of this study is to examine the effect of Self-acupressure application on fatigue and sleep quality in epilepsy patients.

DETAILED DESCRIPTION:
Acupressure is a therapy method performed with an instrument or hand, fingertip, palm, elbow, knee, thumb relaxation and wrist bands on various points representing the waist organs in our body in order to ensure the continuation and balance of the energy in our body.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Volunteering to participate in the research
* Having the ability to use technological tools
* Not having a verbal communication disability (hearing and speaking)
* Not having a diagnosed psychiatric disorder
* Having a scale score of >5 on the Piper Fatigue Scale
* A score of >5 on the Pittsburgh Sleep Quality Scale

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
The Piper Fatigue Scale | At the end of Sessions 1 (each Session 2 days a week)
  It is a 22-item scale that measures four subscales: behavior (6 items), affect (5 items), sensory (5 items), and cognition/mood (6 items). Each item has 11 response categories on a 0-10 metric with verbal descriptors anchoring the endpoints. Each subscale is scored individually and then aggregated together for an overall score, with higher scores reflecting more fatigue.
The Piper Fatigue Scale | At the end of Sessions 16 (each Session 2 days a week)
  It is a 22-item scale that measures four subscales: behavior (6 items), affect (5 items), sensory (5 items), and cognition/mood (6 items). Each item has 11 response categories on a 0-10 metric with verbal descriptors anchoring the endpoints. Each subscale is scored individually and then aggregated together for an overall score, with higher scores reflecting more fatigue.
Pittsburgh Sleep Quality Index (PSQI) | At the end of Sessions 1 (each Session 2 days a week)
  The PSQI is a valid and consistent survey comprising of 19 questions to assess quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients subjective sleep quality, sleep delay, use of sleeping medication and disfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score which is ≤5 indicates "good sleep", and a score which is >5 indicates "poor sleep"
Pittsburgh Sleep Quality Index (PSQI) | At the end of Sessions 16 (each Session 2 days a week)
  The PSQI is a valid and consistent survey comprising of 19 questions to assess quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients subjective sleep quality, sleep delay, use of sleeping medication and disfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score which is ≤5 indicates "good sleep", and a score which is >5 indicates "poor sleep"

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan Bahçecioğlu Turan, PhD, Study Director — Firat University
Locations (1):
- Firat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang T, Zhang Q, Xue X, Yeung A. A systematic review of acupuncture and moxibustion treatment for chronic fatigue syndrome in China. Am J Chin Med. 2008;36(1):1-24. doi: 10.1142/S0192415X08005540. PMID 18306446